CLINICAL TRIAL: NCT02064751
Title: Noninvasive Hemodynamics for MultiPoint(TM) Pacing Programming in Cardiac Resynchronization Therapy Patients
Brief Title: MultiPoint Pacing Programming Guided by Noninvasive Hemodynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD_704
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MultiPoint Pacing (Experimental): CRT with MultiPoint Pacing
  Interventions: Device: CRT with MultiPoint Pacing; Procedure: Hemodynamic measurements for CRT device programming

INTERVENTIONS:
Device: CRT with MultiPoint Pacing
Procedure: Hemodynamic measurements for CRT device programming

SUMMARY:
The purpose of this study is to evaluate noninvasive hemodynamics with MultiPoint™ Pacing (MPP) and biventricular (BiV) pacing under various vector combinations and paced delays in patients receiving cardiac resynchronization therapy (CRT).

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled to undergo de novo implant of a St. Jude Medical CRT-D system
* Be in NYHA II or III functional class with approved standard indication by ESC/EHRA Guidelines
* Have the ability to provide informed consent for study participation and be willing and able to comply with the Clinical Investigation Plan (CIP) described evaluations and follow-up schedule

Exclusion Criteria:

* Have persistent or permanent atrial fibrillation
* Have a recent myocardial infarction within 40 days prior to enrollment
* Have undergone cardiac surgery or coronary revascularization procedure within 3 months prior to enrollment or be scheduled for such procedures in the following 12 months
* Have had a recent Cerebrovascular Accident (CVA) or Transient Ischemic Attack (TIA) within 3 months prior to enrollment
* Have had intravenous inotropic support in the last 30 days
* Be scheduled or considered for heart transplantation over the next 12 months
* Be less than 18 years of age
* Be pregnant or plan to become pregnant over the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure changes in hemodynamics during BiV pacing and MPP | up to 6-months

SECONDARY OUTCOMES:
echocardiographic changes to MPP programming guided by noninvasive hemodynamic measurements | 6 months
  End systolic volume will be assessed at 6-month follow-up visit and compared to that of baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Leclercq, MD, PhD, Principal Investigator — University Hospital Rennes, Rennes, France
Locations (4):
- Medizinische Universität Graz, Graz, Austria
- CHU Rennes, Rennes, France
- Italy (2):
  - Niguarda Hospital, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia